CLINICAL TRIAL: NCT04689113
Title: The Effect of Incontinence Health Belief Development Program on Women's Urinary Incontinence Awareness and Health Beliefs
Brief Title: The Effect of Program on Women's Urinary Incontinence Awareness and Health Beliefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ilknur Aydin Avci, Head of Nursing Department, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ODM.0.20.08/111-224
Record Dates: First submitted 2020-12-09; First posted 2020-12-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Urinary Incontinence
Keywords: kegel exercise; urinary incontinence; Awareness; Health Belief Model; Training; Randomization
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): ıntervention group After determining the women according to the research criteria, they were randomized into intervention and control groups.Firstly, Pre-tests were applied to the women in the experimental group. The Incontinence Health Belief Development Program was applied to the women in the experimental group as 5 sessions.This program includes the following topics; urinary system anatomy and physiology, urinary incontinence and risk factors, definition of kegel exercise and its place in urinary incontinence treatment, kegel exercise applied expression, health motivation. A WhatsApp group was established to remind women in the intervention group about the kegel exercise 3 times a day for 3 months to increase their self-efficacy. In addition, a facebook group was opened and posts about urinary incontinence and kegel exercises were made. Posttests were made 3 months after the training ended
  Interventions: Behavioral: Incontinence Health Belief Development Program
- Control Group (No Intervention): Firstly, Pre-tests were applied to the women in the control group. No intervention was applied to this group.Posttests were made 3 months after pre-test.

INTERVENTIONS:
Behavioral: Incontinence Health Belief Development Program — After the applied interventions, it is desired to develop kegel exercise behavior in women.
  Arms: Intervention Group

SUMMARY:
Background: The aim of this study is to determine the effect of "Incontinence Health Belief Development Program" on urinary incontinence awareness and health beliefs of women in premenopausal period.The research was conducted in a randomized controlled double-blind pretest-posttest control group experimental research design type.The data of the research were collected in Samsun / Atakum District Healthy Life Center and three Family Health Centers. The study was completed with 76 women in the experimental group and 77 women in the control group. The pre-test data of the study were collected using the sociodemographic characteristics information form , the Incontinence Awareness Scale (ISI), the "Health Belief Scale for Urinary Incontinence and Kegel Exercise" and the "Broome Pelvic Muscle Self-Efficacy Scale" for the experimental and control groups.A 5-week "Incontinence Health Belief Development Program" was applied to the experimental group. Posttests were applied to the experimental and control groups 3 months after the program. Descriptive statistics, paired t test, chi-square, Mann-Whitney U, Wilcoxon analysis were used in the analysis of the data.

What does this paper contribute?

*Urinary incontinence awareness, health belief on urinary incontinence and kegel exercise and pelvic muscle self-efficacy of women increased after the Incontinence Health Belief Development Program based on the health belief model.

DETAILED DESCRIPTION:
Aim of study The aim of this study is to determine the effect of "Incontinence Health Belief Development Program" on urinary incontinence awareness and health beliefs of women in premenopausal period.

Study design ans setting The research was conducted in a randomized controlled double-blind pretest-posttest control group experimental research design type. To avoid bias the participants were not told whether they were in the experimental or the control group. The randomized clinical trial was based on the guidelines proposed by the Consolidated standard of Reporting Trials- CONSORT 2010. The data of the research were collected in Samsun / Atakum District Healthy Life Center and three Family Health Centers between November 2019- September 2020.

Randomization An intervention group and a control group formed using the research randomizer software. the program used random numbers to select participants and randomly assign them to the experimental or control group(total 160 women, each group 80 women).

Blinding of data collectors and statistician was implemented in this randomized blinded study. another researcher who did not know the group assignments coded the data in the computer. after statistical analysis was conducted and research report was written, assistant researcher explained tge codes for experimental and control group. Therefore, blinding of the collectors, statistical analysis and report writing was provided.

Implementing the Incontinence Health Belief Development Program The trainings were applied to the women in the experimental group in groups of 10 in the Atakum Healthy Life Center in 5 sessions of 45-60 minutes and 5 weeks. For 5 weeks, 8 group trainings were conducted by taking two different groups every week, 4 days a week. Also Establishing Whatsapp and Facebook Groups A WhatsApp group was established to remind women in the intervention group about the kegel exercise 3 times a day for 3 months to increase their self-efficacy. In addition, a facebook group was opened and posts about urinary incontinence and kegel exercises were made.

Data Collection Tools The pre-test data of the study were collected using the sociodemographic characteristics information form , the Incontinence Awareness Scale (ISI), the "Health Belief Scale for Urinary Incontinence and Kegel Exercise" and the "Broome Pelvic Muscle Self-Efficacy Scale" for the experimental and control groups.

Introductory Question Form: Introductory question form was developed by the researcher and consists of questions involving sociodemographic characteristics, gynecological features and urinary incontinence and kegel exercise of people (age, gender, marital status, education status, etc.).

Incontinence Awareness Scale: The urinary incontinence awareness scale, developed by Avci et al. (2017) to measure individuals' awareness of urinary incontinence, consists of 26 items. It consists of 5 sub-dimensions: factors that prevent it from being accepted as a health problem, coping with urinary incontinence, health motivation, restriction and fear of urinary incontinence. Scores obtained from sub-dimensions; For the factors preventing its acceptance as a health problem sub-dimension, min 8, max 40; For health motivation sub-dimension, min 5, max 25; For the sub-dimension of dealing with urinary incontinence, min 6, max 30; For restriction sub-dimension min 3, max 15; For the subscale for fear of urinary incontinence, the minimum is 4 and the maximum is 20. The scale does not have a total score.Having a high score in the factors preventing its acceptance as a health problem indicates that it accepts urinary incontinence as a health problem.High scores on the sub-dimensions of restriction and incontinence indicate that he does not have a fear of restriction and urinary incontinence.Low scores on the health motivation and coping with urinary incontinence sub-dimensions indicate that their health motivation and coping with urinary incontinence are better.

Health Belief Scale for Urinary Incontinence and Kegel Exercise: The scale developed by Avcı and Yıldırım (2019) based on the health belief model to determine the beliefs of individuals about urinary incontinence and kegel exercise, consists of 49 questions in 5-point likert type. Scale items are separated according to susceptibility, seriousness, health motivation, Kegel exercise benefit perception, Kegel exercise barrier perception and self-efficacy subdimensions created according to health belief model. Responses given to each statement in the scale are in 5-point Likert type and all statements are positive. Scores obtained from subdimensions vary between 9-45 for susceptibility subdimension; between 14-70 for seriousness subdimension; between 5-25 for health motivation subdimension; between 7-35 for Kegel exercise benefit perception subdimension; between 9-45 Kegel exercise barrier perception subdimension and between 5-25 for self-efficacy subdimension. There is no total score of the scale. Increasing scores indicate positive perception for susceptibility, seriousness, health motivation, Kegel exercise benefit perception and self-efficacy subdimensions and negative perception for Kegel exercise barrier perception. Increasing scores mean that susceptibility, seriousness and motivation increase; that benefits are perceived high for benefit perception while barriers are perceived high for barrier perception. Cronbach's alphas in the validity and reliability study of the scale are as follows for the sub-dimensions: sensitivity: 0.89; severity: 0.91; health motivation: 0.79; kegel exercise benefit perception: 0.94; kegel exercise barrier perception: 0,90; self-efficacy: 0.89.

Broome Pelvic Muscle Self-Efficacy Scale: Developed by Broome (1999) to measure the perception of self-efficacy in pelvic floor muscle exercise practice and to provide clinicians with a valid and reliable measurement tool in pelvic floor muscle exercise, the scale was validated in Turkish by Zengin and Pınar in 2012. The scale, which consists of 23 statements in total, consists of two sub-dimensions: "effectiveness expectation" and "result expectation". Total scale score is determined by taking the average of the scores obtained from all expressions in the scale. The sub-dimension score is calculated by the average of the total score of the expressions of that dimension. The total score of the scale varies between 0-100; A score of 32 or less indicates low self-efficacy, 33-66 points medium, and a score above 66 indicates high self-efficacy. The validity and reliability of the scale is Cronbach's alpha: 0.95.

Evaluation of Data SPSS 23.0 statistical package program (Statistical Package for the Social Sciences, Chicago, Illinois) was used for statistical analysis and evaluation of the data. Whether the data showed normal distribution was checked with the Kolmogorov-Smirnov test. Independent samples t test and Mann Whitney U test were used to compare data between groups according to normality test. Paired samples t test and Wilcoxon test were used to compare the pre-test and post-test values within the group. The Chi-square test and two ratio tests were used to analyze categorical data. Significance level was taken as p <.05.

Research Budget:

Financial support of the research provided by the Scientific and Technological Research Council of Turkey (TUBITAK) 1002 Short-term Support Program (issue number 219S160).

Ethical aspects: Study approval was given by Ondokuz Mayıs University Clinical Research Ethics Committee. (Decision No: B.30.2.ODM.0.20.08 / 111-224). All participants were informed about tis study and obtained orat-written informed consents.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman over the age of 45 in the premenopausal period who has not entered menopause
* Being able to communicate and volunteer
* Not having urinary incontinence
* Absence of a disease affecting the genital and urinary system (based on self-report)
* Using a smart mobile phone (to be included in Facebook and whatsapp groups)
* There is no obstacle to doing Kegel exercise

Exclusion Criteria:

* Having entered the menopause period
* Refusing to participate in research
* Having a problem with the genito-urinary system Previous treatment for urinary incontinence
* Not having a smart mobile phone
* Not using Facebook and Whatsapp Having urinary incontinence

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since the prevalence of urinary incontinence increases during menopause, only women in the premenopausal period were recruited.
Enrollment: 160 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Incontinence Awareness Scale | 3 month
  The urinary incontinence awareness scale, developed by Avci et al. (2017) to measure individuals' awareness of urinary incontinence, consists of 26 items. It consists of 5 sub-dimensions: factors that prevent it from being accepted as a health problem, coping with urinary incontinence, health motivation, restriction and fear of urinary incontinence. The scale does not have a total score.Having a high score in the factors preventing its acceptance as a health problem indicates that it accepts urinary incontinence as a health problem.High scores on the sub-dimensions of restriction and incontinence indicate that he does not have a fear of restriction and urinary incontinence.Low scores on the health motivation and coping with urinary incontinence sub-dimensions indicate that their health motivation and coping with urinary incontinence are betterence.
Health Belief Scale for Urinary Incontinence and Kegel Exercise | 3 month
  The scale consists of 49 questions in 5-point likert type. Scale items are separated according to susceptibility, seriousness, health motivation, Kegel exercise benefit perception, Kegel exercise barrier perception and self-efficacy subdimensions created according to health belief model. There is no total score of the scale. Increasing scores indicate positive perception for susceptibility, seriousness, health motivation, Kegel exercise benefit perception and self-efficacy subdimensions and negative perception for Kegel exercise barrier perception. Increasing scores mean that susceptibility, seriousness and motivation increase; that benefits are perceived high for benefit perception while barriers are perceived high for barrier perception.
Broome Pelvic Muscle Self-Efficacy Scale | 3 month
  The scale, which consists of 23 statements in total, consists of two sub-dimensions: "effectiveness expectation" and "result expectation". Total scale score is determined by taking the average of the scores obtained from all expressions in the scale. The sub-dimension score is calculated by the average of the total score of the expressions of that dimension. The total score of the scale varies between 0-100; A score of 32 or less indicates low self-efficacy, 33-66 points medium, and a score above 66 indicates high self-efficacy. The validity and reliability of the scale is Cronbach's alpha: 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Aydin AVCİ, Prof, Study Director — Ondokuz Mayıs University; Yakup BOSTANCI, Assoc.Prof., Study Chair — Ondokuz Mayıs University; Eren Yıldırım, Dr., Study Chair — Liv Hospital Samsun
Locations (1):
- Liv Hospital Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to [restrictions e.g. their containing information that could compromise the privacy of research participants].